CLINICAL TRIAL: NCT05217264
Title: Reliability and Validity of the Turkish Version of the High Activity Arthroplasty Score
Brief Title: Adaptation of High Activity Arthroplasty Score to Turkish
Status: Completed | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Zeynal Yasacı, Research Assistant, Harran University
Other Study IDs: Observational
Record Dates: First submitted 2022-01-18; First posted 2022-02-01 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Arthropathy; Surgery--Complications; Physical Disability
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assesment — This is a single-center, prospective, observational study. The assessment and reporting will be followed the Consensus-Based Standards for the Selection of Health Status Measurement Instruments (COSMIN) checklist.

SUMMARY:
The objectives of this study were the translation, cross-cultural adaptation, and assessment of the psychometric properties of the Turkish High-Activity Arthroplasty Score (HAAS) in patients with primary TKA.

DETAILED DESCRIPTION:
The purpose of this study is to translate and cross-culturally adapt the HAAS instrument into Turkish and investigate its psychometric properties. For cross-cultural adaptation, two bi-lingual translators used the back-translation procedure. Within a 5-to-7-day period after the first assessment, the participants will complete the Turkish version of HAAS to evaluate test-retest reliability. Cronbach's alpha (α) will use to assess internal consistency. The correlations with the Turkish version of the KOOS, SF-36 and FJS-12 will determine to check the validity.

ELIGIBILITY:
Inclusion Criteria:

1. Primary THA/TKA due to primary osteoarthritis for >6 months,
2. Age <65
3. To be able to communicate in Turkish
4. Agree to participate in the study

Exclusion Criteria:

1. who do not agree to participate in the study 2- who will undergo 2nd revision TKA 3- who have undergone lower extremity surgery and thus have sequelae 4-having cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with a total or unicompartmental knee prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
High-Activity Arthroplasty Score | Baseline,
  The HAAS questionnaire, developed in 2010, is self-reported and comprises the four items walking, running, stair climbing, and the activity level [20]. The response level for each item ranges from normal function to serious limitation. The patient selects the highest possible level of his functional ability for each item. A point system for each item is applied whereby a higher score indicates a higher functional ability. The total score ranges from 0 to 18 points. The original version provides no instruction regarding missing answers.

SECONDARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of a knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). A Likert scale is used, and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems
SF-36 | Baseline
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study. It comprises 36 questions which cover eight domains of health:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions
Forgotten Joint Score | Baseline
  The FJS-12 was developed to identify the awareness of an artificial joint (hip or knee) during activities of daily living. It uses a 5-point Likert response format (0, never; 1, almost; 2, seldom; 3, sometimes; and 4, mostly) consisting of 12 items that assess "the patient's ability to forget the artificial joint in everyday life" following activities of daily living -in bed at night; sitting in a chair (>1hr); walking (>15 min); taking bath; traveling in a car; climbing stairs; walking on uneven ground; standing up from a low sitting position; standing for long periods; doing housework or gardening; taking a walk or hiking, and involving in a sports activity. The raw scores are transformed to range from 0 to 100 points. High scores indicate a good outcome, which means a high degree of "forgetting" the joint.
High-Activity Arthroplasty Score | Within a 3-to-5-day period after the first assessment (Second assessment)
  The HAAS questionnaire, developed in 2010, is self-reported and comprises the four items walking, running, stair climbing, and the activity level [20]. The response level for each item ranges from normal function to serious limitation. The patient selects the highest possible level of his functional ability for each item. A point system for each item is applied whereby a higher score indicates a higher functional ability. The total score ranges from 0 to 18 points. The original version provides no instruction regarding missing answers.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynal YASACI, MSc, Principal Investigator — Harran University
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)